CLINICAL TRIAL: NCT01341262
Title: Thalidomide-Dexamethasone Incorporated Into Double Autologous Stem-Cell Transplantation for Patients Less Than 65 Years of Age With Newly Diagnosed Multiple Myeloma
Brief Title: THAL-DEX Incorporated Into Double PBSC Autotransplantation for Untreated Multiple Myeloma (MM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Prof. Michele Cavo, Azienda Opsedaliera Universitaria di Bologna Policlinico S. Orsola Malpighi
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-BO2002
Record Dates: First submitted 2011-03-31; First posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-03

CONDITIONS: Multiple Myeloma
Keywords: autologous stem cell transplantation; thalidomide; induction therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Dexamethasone; Zoledronic Acid; Cyclophosphamide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Thalidomide — * INDUCTION THERAPY: 100 mg/d on days 1-14, 200 mg/d on days 15-120 (in case of delay of HD-CTX , Thalidomide will be continued until the day before Cyclophosphamide as priming therapy for PBSC collection)
  * AFTER PBSC COLLECTION: 200 mg/d from day after last PBSC collection until the day before first course of MEL-200
  * AFTER FIRST TRANSPLANTATION: 200 mg/d from recovery of hematopoiesis until the day before the second course of MEL-200
Drug: Dexamethasone — * INDUCTION THERAPY: 40 mg/d days 1-4, 9-12 and 17-20 (cycles 1 and 3, 30 days each); 40 mg/d days 1-4 (cycles 2 and 4, 30 days each)
  * AFTER PBSC COLLECTION: 40 mg/d days 1-4 (starting the same day of resumption of Thalidomide)
  * AFTER FIRST TRANSPLANTATION: 40 mg/d days 1-4 (starting the same day of resumption of Thalidomide) for 3 cycles (30 days each)
Drug: Zoledronic acid — * INDUCTION THERAPY: 4 mg i.v. once a cycle for 4 cycles (30 days each)
  * AFTER PBSC COLLECTION: 4 mg i.v. once (the same day of resumption of Thalidomide)
  * AFTER FIRST TRANSPLANTATION: 4 mg i.v. once a cycle (starting the same day of resumption of Thalidomide) for 3 cycles (30 days each)
Drug: Cyclophosphamide — Cyclophosphamide 7 g/sqm + G-CSF 5 mcg/Kg from the day +6 for stem cell mobilisation
Drug: Melphalan — Melphalan 200 mg/sqm on day -1 for first and second ASCT

SUMMARY:
The marked activity of thalidomide (thal) and dexamethasone (dex) in relapsed and refractory multiple myeloma (MM) provided the basis for this phase 2 clinical study aimed at investigating the efficacy and toxicity of thal-dex incorporated into melphalan-based double autologous stem cell transplantation (ASCT)for patients less than 65 years old with newly diagnosed symptomatic MM. Thal-dex was given as primary induction therapy and was then continued throughout the subsequent treatment phases until the day before the second autotransplantation. Primary study endpoints,as evaluated on an intention to treat basis, are response rates to the different treatment phases (induction, first and second ASCT), best response whenever achieved, duration of response (DOR), time to progression (TTP), progression free survival (PFS)and toxicity profile of thal-dex. Secondary endpoints, as evaluated on an intention to treat basis, are overall survival (OS) and clinical outcomes (DOR, TTP, PFS and OS)according to prognostic factors, including cytogenetic abnormalities and imaging features, as detected by 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of symptomatic MM based on standard criteria.
* No prior or current systemic therapy for MM, with exception of steroids.
* At least 18 years and less than 65 years of age.
* Presence of quantifiable M protein in serum or urine.
* Durie & Salmon stage II-III or I with disease progression.
* Adequate organ function (heart, lung).
* No previous deep vein thrombosis and/or recurring thrombophlebitis and/or pulmonary embolisms, confirmed by doppler ultrasound or computed tomography scan.
* Willing and able to comply with the protocol requirements.

Exclusion criteria:

* Diagnosis of smouldering or asymptomatic MM, plasmacell leukemia, solitary plasmocytoma of the bone o extramedullary plasmocytoma.
* Diagnosis of non-secretory MM.
* Prior or current systemic therapy for MM, with exception of steroids.
* More than 65 years of age.
* Female subjects pregnant.
* Non adequate organ function (heart, lung).
* Patient has a prior history of thrombosis or venous thromboembolism or pulmonary embolism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2002-03; Primary Completion 2007-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Response rate (at least PR, VGPR, nCR and CR) to thal-dex induction | 120 days after the start day of tal-dex induction therapy
  Responses are reported by study investigators and centrally reassessed by study coordinator(s). Criteria are those initially proposed by the European Group for Blood and Marrow Transplantation (EBMT), with the addition of nCR (100% M-protein reduction by electrophoresis, but immunofixation-positive)and VGPR (at least 90% reduction of M component).
duration of response (partial response, PR, very good partial response, VGPR, complete response, CR) | Average time period between the day of first achievement of response and the day of first relapse or progression
  Duration of response is calculated from the first achievement of the response (at least PR, at least VGPR, at least CR) to relapse/progression
time to progression (TTP) | Average time period between the start day of induction therapy and the day of relapse or progression
  TTP is calculated from the start date of induction therapy to the date of relapse/progression
progression free survival (PFS) | Average time period between the start day of induction therapy and the day of relapse or progression or death, whichever occurs firstly
  PFS is calculated from the start date of induction therapy to the date of relapse/progression or death for any cause, whichever occurs first
toxicity of thal-dex (induction and subsequent treatment phases) | Within 30 days after the last dose of study drug
  Adverse events are assessed monthly and graded according to the National Cancer Institute Common Toxicity Criteria, version 2. Safety is monitored until 30 days after the last dose of study drug.
Response rate (at least PR, VGPR, nCR and CR) to first ASCT | 90 days after first ASCT
  Responses are reported by study investigators and centrally reassessed by study coordinator(s). Criteria are those initially proposed by the European Group for Blood and Marrow Transplantation (EBMT), with the addition of nCR (100% M-protein reduction by electrophoresis, but immunofixation-positive)and VGPR (at least 90% reduction of M component).
Response rate (at least PR, VGPR, nCR and CR) to second ASCT | 90 days after second ASCT
  Responses are reported by study investigators and centrally reassessed by study coordinator(s). Criteria are those initially proposed by the European Group for Blood and Marrow Transplantation (EBMT), with the addition of nCR (100% M-protein reduction by electrophoresis, but immunofixation-positive)and VGPR (at least 90% reduction of M component).

SECONDARY OUTCOMES:
Overall survival (OS) | Average time period between the start day of induction therapy and the day of death, due to any cause
  OS is measured from the start date of induction therapy until death from any cause
OS by cytogenetic abnormalities | Average time period between the start day of induction therapy and the day of death, due to any cause
  OS is calculated as defined above in patients with or without high risk cytogenetic abnormalities (translocation t(4;14), deletion chromosome 17p, deletion chromosome 13q)
OS by 18F-FDG PET/CT imaging | Average time period between the start day of induction therapy and the day of death, due to any cause
  OS is calculated as defined above in patients with different PET/CT patterns (normal, focal, diffuse, presence or absence of extramedullary disease)
TTP by cytogenetic abnormalities | Average time period between the start day of induction therapy and the day of relapse or progression
  TTP is calculated as defined above in patients with or without high risk cytogenetic abnormalities (translocation t(4;14), deletion chromosome 17p, deletion chromosome 13q)
PFS by cytogenetic abnormalities | Average time period between the start day of induction therapy and the day of relapse or progression or death, whichever occurs firstly
  PFS is calculated as defined above in patients with or without high risk cytogenetic abnormalities (translocation t(4;14), deletion chromosome 17p, deletion chromosome 13q)
TTP by 18F-FDG PET/CT imaging | Average time period between the start day of induction therapy and the day of relapse or progression
  TTP is calculated as defined above in patients with different PET/CT patterns (normal, focal, diffuse, presence or absence of extramedullary disease)
PFS by 18F-FDG PET/CT imaging | Average time period between the start day of induction therapy and the day of relapse or progression or death, whichever occurs firstly
  PFS is calculated as defined above in patients with different PET/CT patterns (normal, focal, diffuse, presence or absence of extramedullary disease)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Cavo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna

REFERENCES:
- [Derived] Zamagni E, Patriarca F, Nanni C, Zannetti B, Englaro E, Pezzi A, Tacchetti P, Buttignol S, Perrone G, Brioli A, Pantani L, Terragna C, Carobolante F, Baccarani M, Fanin R, Fanti S, Cavo M. Prognostic relevance of 18-F FDG PET/CT in newly diagnosed multiple myeloma patients treated with up-front autologous transplantation. Blood. 2011 Dec 1;118(23):5989-95. doi: 10.1182/blood-2011-06-361386. Epub 2011 Sep 6. PMID 21900189